CLINICAL TRIAL: NCT05135637
Title: Integrated Immunization and PHC for Enteric Pathogen Control
Brief Title: Naunehal - Integrated Immunization & MNCH Interventions; A Quasi-Experimental Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Aga Khan University (Other)
Responsible Party: Principal Investigator, Zulfiqar Bhutta, Co-Director, Centre for Global Child Health, The Hospital for Sick Children
Other Study IDs: Naunehal Project
Record Dates: First submitted 2021-11-24; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Under Five Child Health Nutrition and Immunization
Keywords: Maternal & child health, immunization, community engagement
MeSH Terms: interventions — Immunization; Nutritional Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Kharotabad 1 - Intervention Union Council (UC): UC where all interventions (mobile health services, community mobilization, private practitioner engagement and test of Sehat Nishani app) will take place, and the UC will undergo a baseline, midline and endline survey.
  Interventions: Other: Mobile health services; Other: Private practitioner engagement for immunization; Other: Community engagement and mobilization; Other: Sehat Nishani - a health, nutrition and immunization app
- Ward 11 - Control UC: UC where no interventions will be done but the UC will undergo a baseline, midline and endline survey.
- Bhana Mari - Intervention UC: UC where all interventions (mobile health services, community mobilization, private practitioner engagement and test of Sehat Nishani app) will take place, and the UC will undergo a baseline, midline and endline survey.
  Interventions: Other: Mobile health services; Other: Private practitioner engagement for immunization; Other: Community engagement and mobilization; Other: Sehat Nishani - a health, nutrition and immunization app
- Sheikh Junaidabad - Control UC: UC where no interventions will be done but the UC will undergo a baseline, midline and endline survey.
- Bakhmal Ahmedzai - Intervention UC: UC where all interventions (mobile health services, community mobilization, private practitioner engagement and test of Sehat Nishani app) will take place, and the UC will undergo a baseline, midline and endline survey.
  Interventions: Other: Mobile health services; Other: Private practitioner engagement for immunization; Other: Community engagement and mobilization; Other: Sehat Nishani - a health, nutrition and immunization app
- Pahar Khel Thal: UC where no interventions will be done but the UC will undergo a baseline, midline and endline survey.

INTERVENTIONS:
Other: Mobile health services — Mobile health services (MHS) will be deployed with one team per UC. MHS will focus on underserved areas to provide basic health services, immunization, & health and nutrition counseling for under-five children & WRAs.
  Groups: Bakhmal Ahmedzai - Intervention UC; Bhana Mari - Intervention UC; Kharotabad 1 - Intervention Union Council (UC)
Other: Private practitioner engagement for immunization — Private healthcare providers (HCPs) will be taken on board to increase coverage of immunization. HCPs will offer routine vaccination to all under-five children visiting their clinics. Project team will liaison with EPI to arrange vaccines for them.
  Groups: Bakhmal Ahmedzai - Intervention UC; Bhana Mari - Intervention UC; Kharotabad 1 - Intervention Union Council (UC)
Other: Community engagement and mobilization — Community engagement & mobilization will focus on immunization, breastfeeding practices, & optimal care-seeking for both pregnant women and young children. Opinion leaders will be engaged to gain support for activities.
  Groups: Bakhmal Ahmedzai - Intervention UC; Bhana Mari - Intervention UC; Kharotabad 1 - Intervention Union Council (UC)
Other: Sehat Nishani - a health, nutrition and immunization app — Sehat Nishani App will be launched to assess feasibility of a health, & immunization app to capture information on birth, nutrition, immunization & growth records. Lady health workers (LHWs), lady health visitors (LHVs) in government health facilities, EPI vaccinators & HCPs will be engaged to use app.
  Groups: Bakhmal Ahmedzai - Intervention UC; Bhana Mari - Intervention UC; Kharotabad 1 - Intervention Union Council (UC)

SUMMARY:
Maternal, newborn, and child health (MNCH) are an area of concern in Pakistan with many health and nutrition indicators at sub-optimal levels. Although these indicators are slowly improving, the interruption of health and immunization programs due to COVID-19 is projected to have severe impacts on the health of women and children. The purpose of this pilot is to test an integrated strategy of implementing immunization, primary health care, and nutrition services in a high-risk setting of Pakistan.

DETAILED DESCRIPTION:
Study Design: The project will adopt a quasi-experimental prepost study design to assess the impact of the proposed interventions. The three union councils (UCs) are the intervention sites and for each of these target UCs, a separate, matched control UC of comparable size, location and coverage indicators will be identified, with propensity score matching and in consultation with local partners. Baseline and endline surveys will be conducted using the 30x7 techniques. 30 clusters demarcated by the government's polio program from each UC will be randomly selected and 15 households with children under-five selected from each cluster. Thus, to achieve an optimal sample size, 450 households will be surveyed from each of the intervention and control UCs. The survey will focus on household characteristics, immunization coverage, health & care-seeking behaviours, and WASH practices.

Intervention Strategies Naunehal aims to improve health service delivery and enhance uptake, by focusing on four main intervention strategies to be implemented in all three target UCs; community mobilization to enhance awareness and demand, mobile health teams offering MNCH and immunization services, engagement of private sector to increase immunization coverage and testing of a comprehensive health, nutrition, growth, and immunization app, Sehat Nishani. The target group of the project include women of reproductive age (WRA) (15-49 years) and children under-five residing in the UCs.

Community engagement and mobilization will include dissemination of comprehensive messaging on promotion of routine childhood immunization, ideal breastfeeding practices, handwashing, best possible sanitary practices, COVID-prevention, optimal diarrheal management with oral rehydration therapy and zinc supplementation, and appropriate care seeking for both pregnant women and young children. The messages will be communicated via health promotion materials, health awareness sessions, and mosque announcements. Announcements would especially encourage the community for routine childhood immunization and to utilize Naunehal mobile health service, the engaged private practitioners' clinics or government facilities for immunization. An integral step of the community engagement process would be to map and consult with opinion leaders and influential community members, to introduce the project and gain their support for the activities.

Mobile health services (MHS) will be deployed in each of the three pilot UCs, with one team per UC in this pilot phase. Each mobile team will have a female physician, a female vaccinator, and a facilitator and will visit pre-determined areas of the UC daily, for 06 days per week for 12 months. The locations will keep rotating, with an effort to focus on underserved areas where access to and coverage of health facilities is limited. The team will ensure that all COVID-19 -prevention recommendations of the government are followed.

The MHS will provide basic health services, immunization, and health and nutrition counselling targeted towards neonates, young children under-five and WRAs. The services provided by the team are limited to those already approved and recommended by the Pakistan government. Consent will be taken from caregivers and participants so that details on services delivered can be shared and utilized in study analysis. Participants will receive services regardless of whether consent is given or not. Personal identifiers will be removed from data.

The project does not anticipate any major adverse event as routine vaccines are widely used safely. However, guidance will be provided to the team physician on steps to follow in case of an adverse event, including providing emergency medication, stabilization, subsequent referral to a health facility if needed, following up on the child, and directive to return to camp after 24-48 hours for check up. Serious and/or unexpected adverse events will be evaluated and reported to Aga Khan University (AKU) and SickKids. The information on all events will be collected, assessed, and reported on CRFs (Case Report Forms) through routine reporting. If any subject suffers any injury while receiving care, he/she will receive free of cost appropriate care as required and the organization will bear the cost of this care.

Private Sector Engagement is an innovative strategy the project will introduce in the intervention UCs. Naunehal aims to create a replicable model of private sector engagement that can be adopted by the government for long-term sustainability. Private sector healthcare providers (HCPs) including medical practitioners and physicians in the target UCs will be taken on board to increase coverage of routine immunization and improve the quality of maternal and child health services. HCPs will offer age-appropriate routine vaccination, including missed doses, to all under-five children visiting their clinics.

Identification of HCPs will occur during the line listing of the baseline survey, and the engaged HCPs will be trained in collaboration with the District Health Office and the Expanded Programme on Immunization (EPI). Training will primarily focus on immunization of neonates and young children as per the schedule and methods endorsed by EPI. Safety protocols, cold chain maintenance and vaccination recordkeeping will be an integral component of the training program. As well, the HCPs will be trained on use of Naunehal health promotion materials as well as counselling.

Project team will liaison with EPI to arrange vaccines for the private practitioners and supply them on a regular, as-needed basis. The arrangement will ensure that vaccines are ready to be picked up or delivered on a pre-determined day from the EPI office with cold-chain maintenance preparations to the practitioners' clinic. These will include BCG, oral polio vaccine (OPV), injectable polio vaccine (IPV), Pentavalent, Pneumococcal, Measles and Rotavirus vaccines.

An incentive for the practitioners would be that they would receive much promotion and exposure within the UC, during community mobilization and public announcements. As well, it will be an opportunity for them to build linkages with the community and with government partners.

Sehat Nishani App will be launched in the three intervention UCs to assess the feasibility of adopting a birth, health, and immunization app to create a vaccination database and capture information on birth, birth weight, nutrition and growth records essential for follow up of the cohort. Lady health workers (LHWs), lady health visitors (LHVs) in government health facilities, EPI vaccinators and partnering HCPs will be engaged to use the Sehat Nishani app on their existing Android phones.

The health workers will receive the necessary orientation and training to use the app and will receive technical support if needed from the project team. Health workers will have app access via a unique login identity (ID) and password and thus, the app will not be publicly accessible. Data from a single family will be linked via a unique Family ID also accessible via an assigned QR code. While LHWs and HCPs will enter both vaccination and health data for under-two children and WRAs, the vaccinators will only enter vaccination data. Health data for children will include birth history, nutritional history, growth record, and an illness record. For WRAs, in addition to the nutritional and illness history, the app will be designed to record details on antenatal care, delivery and postnatal care. Caregivers would be able to log in to the app with their unique ID number and see their child's record without making any changes or entering any information.

App records will be stored in a cloud-based central database managed by AKU, where child health and nutrition data, vaccinator performance, vaccination rates, children overdue for vaccination, and under-immunized areas can be identified.

Monitoring and Impact Evaluation

Naunehal will undergo rigorous monitoring and evaluation, which will include the following activities. As mentioned, household surveys will be conducted at baseline and at then at the end of the project to assess the impact of interventions.

The Mother & Child Care Trust (MCCT) will conduct an independent monitoring and evaluation of the project. MCCT will track the impact of the project using a range of indicators including the number of births registered, birth dose of OPV and BCG received, receipt rates of pneumococcal conjugate (PCV) and measles vaccine, full immunization rates, and zero dose cases.

A household baseline, midline and endline assessment will be conducted for evaluating coverage of interventions as well as the knowledge, attitude, and practices of the community in the maternal, neonatal and child health (MNCH) and COVID-19 context.

The inclusion criteria for a household would include consent from the family, at least one child less than 5 years of age in the household, and that the family has been living in that particular high-risk UC for at least 6 months (including the child in the household) prior to the day of the interview. However, the household will be eligible even if the only child in household was born in the last six months. Any household where a parent or caregiver is not available to answer questions related to the child's health and immunization, will be excluded. Data collected will be processed and analyzed at the AKU, Karachi.

The surveys will help to develop a comprehensive picture of population distribution, health intervention and immunization coverage for children under-5 years. The baseline will also serve as the basis for targeting and tracking progress. Given the enormous impact that COVID-19 related mitigation strategies have had on routine health services such as antenatal care, childbirth services, immunizations and care seeking, this baseline assessment will also assess bottlenecks and help tailor possible approaches to address these issues.

ELIGIBILITY:
Inclusion Criteria:

* Child, less than five years of age
* Resident of the target union council for at least six months (unless the child was born in the last six months)
* Caretaker/parent give consent to participate

Exclusion Criteria:

* Caretaker/parent has not given consent to participate
* Household has no child less than five years
* Under-five child has moved to union council in past six months

Max Age: 59 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The project will be conducted in Union Council (UC) Bhana Mari (District Peshawar), UC Bakhmal Ahmedzai (District Lakki Marwat) and UC Kharotabad 1 (District Quetta) in Pakistan. The study population is the children under-five in these union councils.
Sampling Method: Non-Probability Sample
Enrollment: 8100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Improve reproductive, maternal, neonatal and child under 5 health services and immunization in selected union councils of Pakistan. | Baseline (February 2021), Midline (November 2021) and Endline (May 2022)

SECONDARY OUTCOMES:
Improved care seeking and health behaviours and utilization of MNCH services, immunization and preventive practices in target communities | Baseline (February 2021), Midline (November 2021) and Endline (May 2022)
Improved and enhanced delivery of integrated immunization and health services for women, and children under five in the target UCs. | Baseline (February 2021), Midline (November 2021) and Endline (May 2022)

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar Bhutta, Principal Investigator — SickKids Centre for Global Child Health
Locations (1):
- Trust for Vaccines and Immunization, Karachi, Pakistan

REFERENCES:
- [Derived] Ataullahjan A, Khan A, Islam M, Tahir R, Anwar S, Ahmed I, Nauman A, Bhutta ZA. NAUNEHAL; Integrated immunization and MNCH interventions: A quasi-experimental study-Protocol. PLoS One. 2023 Jun 29;18(6):e0287722. doi: 10.1371/journal.pone.0287722. eCollection 2023. PMID 37384671